CLINICAL TRIAL: NCT07107659
Title: Safety and Efficacy of ONTO1 in Lupus
Brief Title: Safety and Efficacy of ONT01 in Lupus
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Principal Investigator, Timothy Niewold, Principal Investigator, Hospital for Special Surgery, New York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0364
Record Dates: First submitted 2025-07-08; First posted 2025-08-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Lupus Nephritis (LN); Lupus Nephritis - WHO Class III; Lupus Nephritis - WHO Class IV; Lupus Nephritis - World Health Organization (WHO) Class III; Lupus; SLE; Systemic Lupus Erythematosus; Systemic Lupus Erythematosus (Disorder)
Keywords: Lupus Nephritis; Lupus; SLE
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- This study will treat patients with Lupus Nephritis (LN) or Systemic Lupus Erythematosus (SLE). (Experimental): Lupus Nephritis
  Interventions: Drug: ONT01 is a small molecule CD11b modulator.

INTERVENTIONS:
Drug: ONT01 is a small molecule CD11b modulator. — ONT01 will be administered orally twice daily (in the morning and in the evening at approximately 12 hours apart and approximately the same time each day) and should be taken as whole tablets (not crushed) under fasted conditions (2 hours before and 1 hour after each dose) with 8 oz/240 mL of water.

SUMMARY:
ONT01 is a drug that is being studied for the treatment of Lupus Nephritis (LN) and Systemic Lupus Erythematosus (SLE) and is not approved by the FDA. The purpose of this study is to better determine whether ONT01 is safe and tolerated by people with lupus nephritis or SLE. The study also looks at how the administration of ONT01 in combination with widely used treatments given for lupus, including the medication mycophenolate mofetil and others, can improve symptoms of lupus. A total of 61 participants will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old and able to provide informed consent to participate.
2. Diagnosis of SLE and have fulfilled the ACR classification criteria for SLE during the course of their disease.
3. Active non-renal SLE, with one active non-renal clinical manifestation, who have failed at least 1 disease modifying anti-rheumatic drug (DMARD) therapy (not including hydroxychloroquine and corticosteroids)

   * Active non-renal SLE is defined as having a SLEDAI of 6 or greater (with at least 1 non-renal clinical domain) OR Active nephritis defined as having a no or partial response after initial induction and maintenance therapy with mycophenolate mofetil (and other standard of care therapies) for 3 months or more for class III, IV, IV, V (or combination) nephritis.
   * Active LN is defined as follows: a. kidney biopsy showing Class III, IV, V, III+V, or IV+V, within 1 year from screening, AND b. 24-hour urine protein/creatinine ratio >=1g/g at screening, AND c. absence of partial renal response (PRR)
   * Partial renal response (PRR) is defined as a. 24-hour UPCR improved by >=25% after 3 months from the start of induction standard of care (SOC) therapy (baseline), or >= 50% after 6 months from the induction therapy (UPCR), AND b. 24-hour UPCR<2g/g if baseline was < 3g/g, OR < 3g/g if baseline at induction was >= 3g/g. AND d. EGFR>=60 ml/min/1.73 M2 or no less than 80% of Baseline eGFR (at induction) AND e. No intercurrent rescue therapy, death, or early SOC treatment discontinuation or study withdrawal No response (NR) is defined as a. no achievement of at least a partial renal response, OR b. use of intercurrent rescue therapy, OR c. death
4. Female patients who are women of childbearing potential must agree to use a highly effective form of contraception during the study and for at least 120 days after last exposure to study drug. Male patients with female partners of childbearing potential must use effective barrier contraception (i.e., condoms) during the study and for at least 120 days after last exposure to study drug. Also, patients may not proceed with sperm or egg donation during the study and for at least 120 days after the last exposure to study drug

Exclusion Criteria:

1. Any condition, including any uncontrolled disease (eg, asthma, interstitial lung disease, pulmonary arterial hypertension, morbid obesity), that in the Sponsor-Investigator's opinion constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation.
2. Active central nervous system SLE associated with significant cognitive impairment leading to inability to provide informed consent and/or comply with the protocol.
3. Comorbidities requiring systemic corticosteroid (CS) therapy, such as asthma or inflammatory bowel disease. Systemic is defined as oral, rectal or any injectable route of administration (thus stable dosing by other routes is allowed, including inhaled, topical, ophthalmic, otic, and intranasal).
4. Active clinically significant viral, bacterial or fungal infection, or any major episode of infection requiring hospitalization or treatment with parenteral anti-infectives within 4 weeks of or during the Screening Visit, or completion of oral anti-infectives within 2 weeks before or during the Screening Visit.
5. History of positive human immunodeficiency virus (HIV), hepatitis C antibody and/or polymerase chain reaction, hepatitis B surface antigen (HBsAg) (+), and/or hepatitis B core IgG and/or IgM antibody (+) at the Screening Visit.
6. History, or current diagnosis, of active tuberculosis (TB), or untreated latent TB infection (LTBI), determined by a positive QuantiFERON test at the Screening Visit
7. History of malignancy (hematologic or solid tumor) within 10 years prior to Screening Visit, except adequately treated basal cell or squamous cell carcinomas of the skin (no more than 3 lesions requiring treatment in lifetime) or adequately treated carcinoma in situ/cervical intraepithelial neoplasia of the uterine cervix.
8. Immunization with live or live-attenuated vaccines within 1 month before or during the Screening period.
9. Initiation of, or change in, dosing of an angiotensin-converting enzyme inhibitor or angiotensin receptor blocker within 2 weeks before the Screening Visit or during the Screening period.
10. Treatment with Voclosporin or Cyclophosphamide at time of screening.
11. Treatment with other investigational agents within the last 3 months or 5 half-lives, or as per washout requirement from the previous protocol, whichever is longest, prior to the Screening Visit.
12. Clinically significant abnormalities in laboratory tests, unless attributable to active SLE at the Screening Visit

    * Aspartate aminotransferase, alanine aminotransferase or alkaline phosphatase level > 2.5 × upper limit of normal (ULN), or
    * Total bilirubin > 1.5 × ULN, or
    * Hemoglobin < 5.0 mmol/L [9 g/dL], or
    * White blood cells < 2.5 × 109/L, or
    * Absolute neutrophil count < 1500 /mm3, or
    * Platelets < 75 × 109/L
13. Clinically significant chest imaging (e.g. X-ray, computed tomography or magnetic resonance imaging [MRI]) abnormalities per Sponsor-Investigator opinion (e.g. interstitial lung disease) or evidence of active TB on chest X-ray. Chest imaging study must have been performed in 3 months prior to the Screening Visit or during the Screening period.
14. Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
15. Patients are unable or unwilling to adhere to the contraception requirements outlined in inclusion criteria 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2026-09-04 (Estimated); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events, Study Completion versus Withdrawal | From Enrollment until 18 weeks
  This pilot phase 1 study will establish the highest safe dose of ONT01 and help generate preliminary evidence in support of future, large-scale, multi-site, controlled Phase 2 efficacy clinical trials with ONT01 in lupus, so that it can be developed as a novel, myeloid directed, oral therapeutic for lupus.

SECONDARY OUTCOMES:
Effect on SLE and Lupus Nephritis Biomarkers at Day 28 | From baseline until Day 28
  Proportion of patients with statistically significant reduction in
  * suPAR (ng/mL)
  * Proteinuria (protein to creatinine ratio (mg/g)
  * C5a (ng/mL)
  * IL-16 (ng/mL)
  * Anti-dsDNA antibodies (IU/mL)
  * Active SLE symptoms (presence or absence of active symptoms as defined by the SLEDAI criteria)
  Lupus Nephritis secondary outcomes: 25 participants will be enrolled. which will allow us to detect a 1.24-fold difference in a biomarker with 80% power, assuming a 30% standard deviation, with an alpha of 0.01.
  Active non-renal lupus secondary outcomes: 36 participants will be enrolled, which will allow us to detect a 1.24-fold difference in a biomarker with 80% power, assuming 30% standard deviation, with an alpha of 0.01.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No